CLINICAL TRIAL: NCT01972243
Title: Identification of Patients at Low Risk of Recurrent Venous Thromboembolism After Stopping Anticoagulant Treatment: A Prospective Multicenter Cohort Study (Validation of the Vienna Prediction Model)
Brief Title: Risk of Recurrent Venous Thrombosis: A Validation Study of the Vienna Prediction Model
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sabine Eichinger, MD, Medical University of Vienna
Other Study IDs: KLI316
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Venous Thromboembolism
Keywords: risk of recurrent
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- venous thromboembolism
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Because of a high recurrence risk after unprovoked venous thromboembolism (VTE) indefinite anticoagulation is recommended, but confers a considerable bleeding risk. It is important to identify patients, in whom the recurrence risk is lower than the expected bleeding risk, and who will not benefit from long term anticoagulation. By use of a scoring model (Vienna Prediction Model), patients can be stratified according to their recurrence risk based on their sex, location of VTE and D-Dimer. Before implementation in routine care, an independent validation is required. Patients with unprovoked VTE will stop anticoagulation after 3-7 months and the recurrence risk will be estimated by use of the Vienna Prediction Model. Low risk patients with a score of <180 will be included and will be left untreated. Patients with a high score will not be included and their management will follow current guidelines. Follow-up will be two years and the endpoint will be recurrent symptomatic VTE.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years symptomatic uni- or bilateral proximal (including the trifurcation area, popliteal, superficial femoral, deep femoral, common femoral and iliac vein) or distal DVT of the leg and/or symptomatic PE.

VTE not provoked by one of the following temporary risk factors: surgery, trauma,pregnancy, cancer, immobilisation.

Exclusion Criteria:

History of previous VTE; anticoagulation for longer than 6 months; reasons for long-term anticoagulation other than VTE; poor patient compliance; no consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: first unprovoked deep vein thrombosis or pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2013-09; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
recurrent venous thromboembolism | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria